CLINICAL TRIAL: NCT00514891
Title: Evaluation of the Impact on Mortality and Morbidity of the WHO Recommended Vitamin A Supplementation at First Immunisation Contact After 6 Months of Age
Brief Title: Impact of the WHO Recommended Vitamin A Supplementation at Immunisation Contacts
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Reccomended by DSMB after review of planned interim analyses.
Sponsor: Bandim Health Project (Other)
Collaborators: Ministry of Health, Guinea-Bissau (Unknown); University of Aarhus (Other)
Responsible Party: Ane Fisker, Bandim Health Project
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CVK-2006-7041-99
Record Dates: First submitted 2007-08-08; First posted 2007-08-10 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-01

CONDITIONS: Mortality; Morbidity
MeSH Terms: interventions — Vitamin A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Vitamin A supplementation
  Interventions: Biological: Vitamin A
- 2 (Placebo Comparator): Placebo
  Interventions: Biological: Vitamin A

INTERVENTIONS:
Biological: Vitamin A — The effect of vitamin A given with different vaccines will be studied

SUMMARY:
High-dose vitamin A to children above 6 months of age reduces all-cause mortality by 23-30%. The WHO recommends vitamin A supplementation (VAS) with the first vaccine after 6 months of age. However, the effect of providing VAS with vaccines has never been investigated. We have hypothesised that the effect of VAS depends on the immune stimulus at the time of supplementation. Hence, the effect might vary depending on which type of vaccine it is given with. In particular, we hypothesised that VAS might be beneficial when given with measles vaccine but not when given with DTP vaccine. Normally the first vaccine after 6 months of age would be a measles vaccine, but many children come late for their DTP vaccinations and receive DTP alone or together with measles vaccine. Hence, it is important to study whether the effect of VAS is the same irrespective of the vaccine(s) administered at the same time.

Guinea-Bissau has not yet implemented the WHO vitamin A policy of providing VAS with vaccines, but plans to do so within the next years. Together with the Ministry of Health in Guinea-Bissau, the Bandim Health Project (BHP) in Guinea-Bissau will investigate the effect on mortality and morbidity of implementing the WHO vitamin A policy in Guinea-Bissau. This will be done in a large randomised trial.

BHP has a demographic surveillance system (DSS) which has followed a population of now more than 150,000 individuals for almost 30 years. Children will be randomised to receive VAS or placebo with their first vaccine after 6 months of age, and will be followed through the DSS to assess mortality and morbidity. Based on previous observations, the effects of VAS might differ according to sex and season. The interaction between VAS, sex, and season will also be studied in the present trial. By identifying situations where VAS may be beneficial, ineffective, or even harmful the study may contribute importantly to optimising the VAS policy for low-income countries.

ELIGIBILITY:
Inclusion Criteria:

* Urban area: 6-17-month-old children, presenting for vaccination at a health centre in the study area.
* Rural area: 6-23-month-old children who are missing one or more routine vaccinations when visited by our mobile team.

Exclusion Criteria:

* Normally applied contraindications for receiving vaccinations, including high fever.
* VAS within last month.

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 9500 (Estimated)
Dates: Start 2007-08; Primary Completion 2012-06 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Mortality, morbidity | 1 year

SECONDARY OUTCOMES:
Growth, Vitamin A status, Immunology

CONTACTS AND LOCATIONS:
Overall Officials: Christine S Benn, MD, PhD, Principal Investigator — Bandim Health Project, Statens Serum Institut, Artillerivej 5, 2300 Copenhagen S, Denmark; Peter Aaby, Dr.Med., Study Director — Bandim Health Project, Apartado 861, 1004 Bissau Codex, Guinea-Bissau
Locations (1):
- Bandim Health Project, Apartado 861, Bissau, Guinea-Bissau

REFERENCES:
- [Derived] Fisker AB, Bale C, Rodrigues A, Balde I, Fernandes M, Jorgensen MJ, Danneskiold-Samsoe N, Hornshoj L, Rasmussen J, Christensen ED, Bibby BM, Aaby P, Benn CS. High-dose vitamin A with vaccination after 6 months of age: a randomized trial. Pediatrics. 2014 Sep;134(3):e739-48. doi: 10.1542/peds.2014-0550. PMID 25136048
- [Derived] Fisker AB, Bale C, Jorgensen MJ, Balde I, Hornshoj L, Bibby BM, Aaby P, Benn CS. High-dose vitamin A supplementation administered with vaccinations after 6 months of age: sex-differential adverse reactions and morbidity. Vaccine. 2013 Jun 28;31(31):3191-8. doi: 10.1016/j.vaccine.2013.04.072. Epub 2013 May 14. PMID 23680441
- [Derived] Danneskiold-Samsoe N, Fisker AB, Jorgensen MJ, Ravn H, Andersen A, Balde ID, Leo-Hansen C, Rodrigues A, Aaby P, Benn CS. Determinants of vitamin a deficiency in children between 6 months and 2 years of age in Guinea-Bissau. BMC Public Health. 2013 Feb 25;13:172. doi: 10.1186/1471-2458-13-172. PMID 23442248